CLINICAL TRIAL: NCT02689115
Title: NF-KB1/IKK Epsilon Genetic Expression in Patients With Rheumatoid Arthritis
Brief Title: NFKB1 and IKK Epsilon in Rheumatoid Arthritis
Acronym: NUIRA
Status: Completed | Type: Observational
Sponsor: Asociación Científica Latina A.C. (Other)
Collaborators: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/02
Record Dates: First submitted 2016-02-15; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Nuclear factor Kappa B; IKK epsilon
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clinical activity: Patients with rheumatoid arthritis who met the criteria established by the American College of RheumatologyDisease Activity Score 28 (DAS28) > 3.6.
  Interventions: Other: Genetic relative expression
- Clinical remission: Patients with rheumatoid arthritis with Disease Activity Score 28 (DAS28) < 2.4.
  Interventions: Other: Genetic relative expression

INTERVENTIONS:
Other: Genetic relative expression — The genetic expression of NF-KB1 and IKK epsilon were quantified in both groups.

SUMMARY:
Rheumatoid arthritis (RA) is a systemic and auto-immune disorder whose primary characteristic is the chronic inflammation of joints. The objective of this study was to evaluate whether there was an association between the NF-KB1/IKK epsilon genetic expression and the clinical activity in RA.

60 RA patients were included in the study, 30 with clinical activity and 30 with clinical remission The NF-KB1/IKK epsilon genetic expression was performed by real time quantitative Polymerase chain reaction (qPCR) through the Pfaffl method of relative quantification with Taqman probes.

DETAILED DESCRIPTION:
Patients with a confirmed diagnosis of RA were allocated in two groups based on the Disease Activity Score 28 (DAS28): a) with clinical activity and b) with clinical remission. Key exclusion criteria were patients with any other inflammatory or autoimmune disease and patients with infections. The control group was represented by healthy patients Sample size

The sample size calculation was carried out through the following formula:

n= Nz2 pq /d2(N-1) +z2 pq With N=30, Z=2.46 (99% of confidence), p=0.9, q=0.1, d=0.05 (95% of accuracy). The sample size contained 20 patients with RA.

Anthropometric measurements Weight (kg) and height (m) were calculated in a mechanical column scale (SECA). The patients were classified according to their Body mass index (BMI, weight (Kg)/ height (m)2) as a) normal weight (BMI< 24.9), b) overweight (24.9 kg/m2 <BMI<29.9 kg/m2) and c) obese (BMI> 30 kg/m2).

Lymphocyte extraction Lymphocytes from peripheral blood were extracted using the ACK Lysing Buffer® (Life technologies, Grand Island, NY) kit. Briefly, a venous blood sample in EDTA tube (BD Vacutainer®, Franklin Lakes, NJ), was centrifuged at 3500 rpm during 5-8 minutes. The resulting intermediate white colored phase was extracted and placed in an eppendorf tube; 1 mL of ACK Lysing Buffer® was added and carefully re-suspended. Once again, the suspension was centrifuged at 3500 rpm during 5-8 minutes and the supernatant was discarded. This last step was repeated until the leukocyte package was completely white. Finally, it was added 100 mcl of ACK Lysing Buffer® and frozen at -70ºC for later use.

Genetic expression From the leukocyte package (approximately 10 to 15 mg), it was performed a messenger RNA (mRNA) extraction using the Magna Pure LC RNA isolation kit III (Roche) in the Magna Pure LC 2.0 Instrument. The A260/A280 nm absorbance ratio was >1.8 (quality) and total RNA concentration was calculated by determining absorbance at 260 nm established with the NanoPhotometer (Implen GmbH, Germany) and the extracts were adjusted to a concentration of 20 µg of DNA for the PCR reaction.

Subsequently, the cDNA was synthesized with the Transcriptor High Fidelity cDNA Synthesis Kit (Roche Applied Science). It was performed a real time polymerase chain reaction (qPCR), using the specific primers and probes for NF-KB1, IKK epsilon and 18s (as constitutive gene), using a 7500 Fast Real Time PCR System (Applied Biosystems, Applera UK, Cheshire, UK), mixing TaqMan® Universal PCR Master Mix and the specific probes for each gene NF-KB1 (Hs00765730-m1), IKK epsilon (Hs01063858-m1) and 18S (Hs99999901-s1), (Applied Biosystems, Applera UK, Cheshire, UK).

According to the Ct obtained from the two different groups it was calculated the relative units of expression through the Pfaffl relative quantification method, in which it was used as control a healthy patient.

Statistical analysis The statistical analysis was performed through the Sigmaplot software version 12.0. Parametric and non-parametric test were used in function to the variable distribution: among the parametric test that were performed to compare the groups, the Student´s T-test was included; the non-parametric tests applied were: The Mann-Whitney U test and the Shapiro-Wilk test. Finally, a receiver operating characteristic (ROC) was used for the analysis of the genetic expression of NF-KB1/IKK epsilon with the SPSS software version 22.0.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis criteria established by the American College of Rheumatology (ACR).

Exclusion Criteria:

* Patients with any other inflammatory, autoimmune or neoplastic disease and patients with infections.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The key inclusion criteria were patients with RA who met the criteria established by the American College of Rheumatology (ACR). Two groups were conformed based on the Disease Activity Score 28 (DAS28): a) with clinical activity (DAS28 > 3.6) and b) with clinical remission (DAS28 < 2.4). Key exclusion criteria were patients with any other inflammatory, autoimmune or neoplastic disease and patients with infections. The control group was represented by healthy patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Relative genetic expression of NF-KB1 and IKK epsilon. | Within one month after the patient selection.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD., Study Director — Asociación Científica Latina A.C.

IPD SHARING:
Plan to Share IPD: Undecided